CLINICAL TRIAL: NCT03945058
Title: Effect of Neuromodulation on Inflammation, Endothelial Function and Cognitive Dysfunction in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Neuromodulation of Inflammation and Vascular Function in Systolic Heart Failure
Acronym: TECO-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was unable to meet target enrollment; no results generated.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10410
Record Dates: First submitted 2019-03-15; First posted 2019-05-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Intervention Model Description: This was a pilot study that was terminated. The COVID pandemic prevented the enrollment of more participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Active TVS will be performed by use of a Tragus stimulator device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour daily for 4 weeks.
  Interventions: Device: TVS; Device: SHAM
- CONTROL (Sham Comparator): Sham TVS will be performed by use of a Tragus stimulator device with electrodes attached to the ear lobule. Stimulator will be applied continuously for 1 hour daily for 4weeks.
  Interventions: Device: TVS; Device: SHAM

INTERVENTIONS:
Device: TVS — Active TVS will be performed by use of a Tragus stimulator device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour daily for 4 weeks
Device: SHAM — Active TVS will be performed by use of a Tragus stimulator device with electrodes attached to the earl lobule. Stimulator will be applied continuously for 1 hour daily for 4 weeks.

SUMMARY:
Heart failure (HF) is the leading cause of death in US. It is associated with abnormal vascular function termed endothelial dysfunction. It is also associated with increased stress on the blood vessels and high levels of inflammation. Vagus nerve stimulation can help improve inflammation, vascular function and vascular stress. The investigator has recently completed a study showing that 1 hour of noninvasive vagus stimulation can improve vascular health. However, it is unknown if 4 weeks of stimulation will be beneficial in systolic heart failure.

The purpose of this study is to determine if transcutaneous vagal stimulation (TVS) will lead to improvement in the function of the inner lining of participants' arteries, memory, and in the levels of certain chemical markers of arterial function in the blood.

Participants will be randomized to receive either TVS or a sham stimulation and undergo 4 weeks of stimulation. Vascular function will be assessed by several non-invasive measurements, including Flow Mediate Dilation (FMD), Pulse Wave Analysis (PWA), EndoPAT, and Laser Speckle Contrast Imaging (LSCI). Participants' memory will also be measured through electronic assessments and blood will be collected and analyzed for arterial function chemical markers.

DETAILED DESCRIPTION:
Visit 1: Following tests(to assess vascular function) will be done: 1. FMD 2) LSCI 3) EndoPAT and 4) Pulse wave analysis (PWA). Patients will rest for 10 minutes between each test. They will be trained to use PARASYMTM unit for TVS. Blood collected, serum/plasma will be stored at -80F. Whole blood will be collected in PAXgene tubes. Patients will be instructed to apply TVS to either ear lobule (SHAM) or Tragus(experimental arm). Baseline characteristics will be collected including data on ventricular function(LVEF and left ventricular volumes).

Visit 2 (4 weeks): Follow up tests(FMD,LSCI,EndoPAT,PWA) and repeat blood collection.

Inflammatory cytokines and vascular function assays will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (18 years or older) with Heart failure with reduced ejection fraction (HFrEF), which is a history of symptomatic heart failure with left ventricular ejection fraction (LVEF) of < 40%.

Exclusion Criteria:

1. Patients in overt congestive heart failure / recent acute myocardial infarction (< 3 months) or Unstable angina
2. Active malignancy
3. Pre-menopausal women and post-menopausal women on hormone supplements.
4. Unilateral or bilateral vagotomy
5. Patients with bilateral upper extremity amputation
6. Pregnant patients
7. End-stage renal disease
8. End-stage liver disease
9. History of recurrent vasovagal syncope, Sick sinus syndrome, 2nd- or 3rd-degree atrioventricular (AV) block.
10. Patients with clinically documented upper extremity arterial disease
11. Patients with a body mass index (BMI) >35
12. Significant hypotension (blood pressure <90mmHg) secondary to autonomic dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilation (FMD) | Change in the brachial artery diameter will be compared to baseline change after 4 weeks of TVS or sham.
  FMD is a change in the maximal diameter of the brachial artery. Brachial artery diameter (in millimeters) will be assessed before and after 4 weeks of stimulation using standard ultrasound.
Laser Speckle Contrast Imaging (LSCI) | Change in the perfusion units will be determined at baseline and after 4 weeks of TVS or sham stimulation.
  LSCI based perfusion index and perfusion units will be calculated before and after 4 weeks of TVS or sham stimulation.
EndoPAT | Change in the reactive hyperemia index from baseline and after 4 weeks of TVS or SHAM stimulation
  Hyperemia index measured with ENDOPAT will be calculated before and after 4 weeks of TVS. Hyperemia index will be calculated using the standard ENDOPAT technique using probes placed on bilateral finger.
Pulse Wave Analysis (PWA) | Change in the augmentation index will be calculated at baseline and after 4 weeks of TVS or sham stimulation.
  Arterial elasticity. Augmentation pressure (AP) will be calculated which is expressed as a percentage of the aortic pulse pressure (PP) which is the difference of systolic and diastolic BP(mm Hg).
Biomarkers of inflammation | Change in these biomarkers(% change) over 4 weeks will be calculated.
  Inflammatory cytokines will assayed at baseline and after 4 weeks of stimulation. Cytokines assayed : Il1B,IL-6,IL-17,TNF-a,TGF-b,CRP etc- expressed in pg/ml units).
Biomarkers of endothelial function and oxidative stress | Change in these biomarkers(%) over 4 weeks will be calculated.
  Biomarkers of endothelial function and oxidative stress include: ORAC, HORAC scores expressed as %.

SECONDARY OUTCOMES:
Cognition | Change in the cognition score , as assessed by the CANTAB method will be compared at baseline and after 4 weeks of TVS or sham stimulation.
  Cognition score(%) calculated from Cambridge Neuropsychological Test Automated Battery -CANTAB method . This will be done using a hand held ipad.

CONTACTS AND LOCATIONS:
Overall Officials: Taun Dasari, MD, Principal Investigator — OUHSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No